CLINICAL TRIAL: NCT07163845
Title: Assessment of Chikungunya Virus Seroprevalence Before VLA1553 Vaccination in the Municipalities Selected for Participation in the VLA1553 Pilot Vaccination Strategy in Brazil
Status: Active, not recruiting | Type: Observational
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: Fundação Butantan (Unknown); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Other Study IDs: VLA1553-407
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Live-attenuated CHIKV vaccine VLA1553 — Non-interventional study: VLA1553 is used in the pilot vaccination strategy which is carried out after this observational study.

SUMMARY:
This is a cross-sectional serosurvey using household cluster sampling conducted before the VLA1553 pilot vaccination strategy will be implemented in about 10 municipalities in Brazil.

DETAILED DESCRIPTION:
Households will be selected randomly using a multi-stage random sampling at the census tract, street, and household levels, to select study participants. The study aims to prospectively evaluate the association between vaccination uptake and previous CHIKV exposure (pre-existing immunity to CHIKV infection) in the age-group approved per label in Brazil (e.g., adults [≥18 years of age] or individuals ≥12 years of age). Seroprevalence among vaccinated and unvaccinated individuals will be used to parameterize a probabilistic bias analysis conducted as part of the VE study. Finally, the study will explore the prevalence of CHIKV exposure in the different study communities before the VLA1553 pilot vaccination strategy in individuals ≥2 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals residing in the selected municipalities of Brazil where the VLA1553 pilot vaccination strategy will be implemented.
2. Individuals ≥2 years of age
3. Individuals who sleep 3 nights a week or more in a household that is selected by cluster sampling.

Exclusion Criteria:

1. Individuals or their legally accepted representatives (LAR) who are not willing or not able to provide informed consent (and assent, as required) according to country-specific procedures.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of individuals ≥2 years of age residing in the municipalities where the pilot VLA1553 vaccination strategy will take place and who meet the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 5354 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To prospectively evaluate the association between vaccination uptake and previous CHIKV exposure (pre-existing immunity to CHIKV infection) after implementing a pilot vaccination in the age-group approved per label. | on Day 1

OTHER OUTCOMES:
To evaluate CHIKV seroprevalence in the selected municipalities before the implementation of a pilot vaccination in the population ≥2 years of age | on Day 1
The association, measured as an odds ratio, between vaccination uptake and prevaccination strategy CHIKV seropositivity (IgG) | on Day 1
Pre-vaccination strategy CHIKV seropositivity (IgG) stratified by vaccination status with VLA1553 vaccine, among the population approved per label | on Day 1
Vaccination uptake, measured as cumulative incidence, according to prevaccination strategy CHIKV seropositivity (IgG) | on Day 1
CHIKV seropositivity (IgG) among the study participants ≥2 years of age assessed by rapid diagnostic test (RDT) or Enzyme-Linked Immunosorbent Assay (ELISA) tested on a dried blood spot (DBS) sample before the implementation of the VLA1553 PVS | on Day 1

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Universidade Federal Do Ceará, Fortaleza, Ceará
  - Universidade Federal de Minas Gerais, CT Terapias Avançadas e Inovadoras, Belo Horizonte, Minas Gerais
  - Centro de Pesquisas Clínicas Universidade Federal Sergipe, Hospital e Maternidade São João de Deus, Laranjeiras, Sergipe
  - Fundação Faculdade Regional De Medicina De São José Do Rio Preto, São Pedro, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided